CLINICAL TRIAL: NCT06218797
Title: Effect of Nebulized Dexmedetomidine on Gag Reflex Suppression in Pediatric Upper Gastrointestinal Endoscopy: a Randomized Controlled Trial
Brief Title: Nebulized Dexmedetomidine as a Premedication for Gastrointestinal Endoscopy in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Esra Turunc, Study director, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NDUGIE2023
Record Dates: First submitted 2023-12-27; First posted 2024-01-23 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Pediatric; Sedation
Keywords: Pediatric; Gastrointestinal endoscopy; Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C (Active Comparator): Control group
  Interventions: Other: a routine sedation protocol
- Group ND (Active Comparator): Nebulisation with dexmedetomidine
  Interventions: Drug: Nebulized with dexmedetomidine

INTERVENTIONS:
Other: a routine sedation protocol — In this study group, a routine sedation protocol in our clinic will be applied in the endoscopic unit. Premedication will not be given to the patients.
  Arms: Group C
Drug: Nebulized with dexmedetomidine — Patients will be received nebulisation with dexmedetomidine 2mcg/kg 5 cc 20 minute prior to endoscopy. After that routine sedation protocol in our clinic will be applied.
  Arms: Group ND

SUMMARY:
This study aims to demonstrate that the application of nebulized dexmedetomidine to patients during pediatric upper gastrointestinal endoscopic procedures will significantly reduce the gag reflex and enhance both patient and practitioner comfort

DETAILED DESCRIPTION:
Due to the intolerance of pediatric patients to the insertion of the endoscopic probe during upper gastrointestinal procedures, sedation and analgesia are required. In this patient group, the reflex to vomit is common during probe placement. Discomfort, pain, and hemodynamic changes can occur due to the vomiting reflex. In fact, this situation can lead to serious complications such as esophageal rupture. Inappropriate sedation conditions may result in increased post-procedural pain and agitation in patients.

Therefore, various sedative drugs are used for procedural sedation in pediatric patients. The use of these drugs during gastrointestinal endoscopy in the pediatric population can vary in terms of sedative, hemodynamic, respiratory, and side effects.

Dexmedetomidine, a highly selective alpha-2 agonist with central sedative and anxiolytic properties, has been tested in children for preoperative anxiolysis through nasal and inhalation routes. Due to its bioavailability of up to 82%, it is well absorbed systemically through oral and buccal routes.' It possesses sedative, analgesic, sympatholytic, and hemodynamic stability properties. Even at high doses, it has a unique feature of not causing respiratory depression, which gives it an advantage over other sedatives such as benzodiazepines, opioids, and propofol, all of which can cause dose-dependent respiratory depression. In this regard, it may be a good alternative for procedures like gastrointestinal endoscopy.

Based on these considerations, the investigators plan to conduct a randomized controlled study hypothesizing that nebulized dexmedetomidine as premedication in pediatric patients undergoing gastrointestinal endoscopy will significantly reduce the gag reflex.

108 patients will be included in the study. Patients will be divided into 2 groups.

* The control group (Group C)
* The group receiving nebulized dexmedetomidine (ND) (Group ND).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I and II
* 2 to 17 years of age,
* Patient undergoing in Upper Gastrointestinal Endoscopy

Exclusion Criteria:

* Patients with heart disease
* Patients with mental-motor retardation
* Patients with abnormal upper respiratory tract
* Patients with a history of asthma
* Patients with upper respiratory tract history in the last 4 weeks
* Patients with severe sleep apnea on polysomnography
* ASA >III patients
* Patients with drug allergies

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
gag reflex | through endoscopic procedure up to one hour
  This will be assessed when a vomiting like response will provoked upon introduction of the endoscope.

SECONDARY OUTCOMES:
Endoscopist's level of satisfaction with regard to the occurrence of gagging and the challenges encountered during the procedure | through endoscopic procedure up to one hour
  This will be assessed using an 5-point Likert scale
Depth of sedation | During Procedure (after 1 minute of induction of sedation and allover the time of the procedure every 2 or 3 minutes)
  This will be assessed by Ramsay sedation score
Adverse effects | 2 hours post the procedure
  This will be reported for any adverse effects such as oxygen desaturation, the need for jaw thrust maneuver or manual ventilation, laryngospasm, vomiting, and shivering.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Turunc, Study Director — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayis University, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Turunc E, Ustun YB, Bilgin S, Kaya C, Koksal E, Dost B. Effect of nebulized dexmedetomidine on gag reflex suppression and sedation quality in pediatric patients undergoing gastrointestinal endoscopy: a randomized controlled trial. BMC Anesthesiol. 2025 May 3;25(1):227. doi: 10.1186/s12871-025-03106-x. PMID 40319232